CLINICAL TRIAL: NCT01159444
Title: What do built-in Softwares in Home Ventilators Tell us? An Observational Study of 150 Patients on Home Ventilation
Brief Title: What do built-in Softwares in Home Ventilators Tell us?
Status: Completed | Type: Observational
Sponsor: Ligue Pulmonaire Genevoise (Other)
Responsible Party: Janssens, Jean-Paul, Professor, Division of Pulmonary Diseases/ Geneva University Hospital
Other Study IDs: JPJ/2010
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Ventilation
Keywords: noninvasive ventilation; ventilator software; ventilator settings; domiciliary ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Home bi-level positive pressure ventilators are equipped with built-in softwares which measure and record specific items such as tidal volume, total ventilation, leaks, respiratory rate, cycles triggered by the patient. These items have not to date been described in a large group of patients under home mechanical ventilation.

DETAILED DESCRIPTION:
Observational study of patients under home positive pressure mechanical ventilation, in a stable condition.

Data recorded by ventilator software is downloaded by specialized nurses during elective home visits, as well as spirometry, results of recent pulse oximetry, ventilator settings, diagnosis, and basic anthropometric data.

Items recorded by ventilator software are: tidal volume, total ventilation, apnea and hypopnea index, leaks, percentage of inspiratory cycles triggered by ventilator, spontaneous and back-up respiratory rates.

Results are reported by diagnostic group. Statistical analysis (univariate and multivariate) aims to determine which variables are related to unintentional leaks, and whether ventilator settings differ significantly between diagnostic groups.

ELIGIBILITY:
Inclusion Criteria: - All patients with home noninvasive ventilation with bi-level positive pressure home ventilators with integrated software

Exclusion Criteria:

* Hospitalisation or acute exacerbation;
* Ventilation with a device not equipped with built-in software,
* Ventilation with servo-assisted ventilator
* Invasive ventilation (tracheostomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for at least 3 months in the Geneva Canton Area, followed by the Division of Pulmonary Diseases of Geneva University Hospital, under home ventilation with bi-level positive pressure home ventilators with integrated software for data recording, in stable clinical condition
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2007-02; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Analysis of data downloaded from ventilator software by diagnostic category | one day
  Analysis of data provided by ventilator software during elective home visits by specialized nurses in stable patients under home ventilation. Data includes all ventilator parameters, leaks, tidal volume, total ventilation, respiratory rate, % of cycles triggered by the patient, apnea-hypopnea index, and compliance. Age, gender, BMI, spirometry, type of mask and pulse oximetry are also available. The analysis will describe ventilatory patterns and ventilator settings as a function of diagnosis, as well as factors related to importance of leaks (age, interface, ventilator settings).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, Professor, Principal Investigator — Division of Pulmonary Diseases; Geneva University Hospital
Locations (1):
- Division of Pulmonary Diseases; Geneva University Hospital, Geneva, Canton of Geneva, Switzerland